CLINICAL TRIAL: NCT00505739
Title: Phase II Study of Mifepristone (RU-486) in the Treatment of PR Positive Advanced/Recurrent Endometrioid Adenocarcinoma and Low Grade Endometrial Stromal Sarcoma (LGESS)
Brief Title: Mifepristone for Patients With Endometrial Cancer and LGESS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID01-212
Record Dates: First submitted 2007-07-19; First posted 2007-07-23 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Endometrial Cancer
Keywords: Endometrial Cancer; Low Grade Endometrial Stromal Sarcoma; RU-486; Mifepristone; LGESS
MeSH Terms: conditions — Endometrial Neoplasms; Endometrial Stromal Tumors | interventions — Mifepristone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mifepristone (Experimental)
  Interventions: Drug: Mifepristone

INTERVENTIONS:
Drug: Mifepristone — 200 mg by mouth (PO) Daily x 4 Weeks
  Other Names: RU-486

SUMMARY:
Primary Objectives:

1. To determine the antitumor activity of Mifepristone (RU-486) in patients with advanced or recurrent endometrioid adenocarcinoma or low grade endometrial stromal sarcoma (LGESS).
2. To evaluate the quantitative and qualitative toxicities of Mifepristone in this patient population.
3. To evaluate at a tissue level the effect of Mifepristone on estrogen and progesterone receptors post treatment and to evaluate other markers that may reflect effects of Mifepristone on cancer cell growth.
4. To evaluate the effect of the agent and dosing schedule on the patient's quality of life.

DETAILED DESCRIPTION:
Mifepristone is a drug that has been approved for use in the termination of pregnancy. It has been studied in women with breast and ovarian cancer.

Before treatment starts, patients will have a complete checkup, blood tests, a CT scan, and a chest x-ray. Women able to have children must have a negative urine pregnancy test. Blood tests and a complete checkup will also be done within 3 days of starting each course of therapy and a month after treatment ends. Tumors will be measured by CT scans once every 2-3 months and at the end of treatment.

Patients in this study will take Mifepristone in the form of a pill by mouth every day. Each course of therapy is 4 weeks long. Patients will see their doctor for an exam and blood tests before they begin each 4 week course of therapy. The dose of Mifepristone may be lowered if the patient has side effects. Patients who have a complete response (there is no evidence of cancer by physical exam or x-ray) will continue taking Mifepristone for 2 years after this response is documented. Other patients will take Mifepristone for as long as it benefits them.

This is an investigational study. At least 12 and as many as 37 patients will take part in this study. Patients from MD Anderson Cancer Center and Gynecologic Oncology of Houston, P.A. will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic diagnosis of advanced/recurrent endometrioid adenocarcinoma or low grade endometrial stromal sarcoma (LGESS) not amenable to curative surgery or radiotherapy.
2. Patients should have previously undergone radical surgery (minimum of total abdominal hysterectomy and bilateral salpingoophorectomy) definitive radiation therapy, or not be candidates for such procedures.
3. The primary (including archived specimens) or recurrent tumor must be PR positive. Hormone receptor positivity is defined as PR positivity in >/+10% cells by immunohistochemistry.
4. Prior radiotherapy must have been completed at least 2 weeks prior to the initiation of Mifepristone and patients must have recovered from the acute side effects of such treatment.
5. Performance status < Zubrod 2.
6. Estimated life expectancy of at least 12 weeks.
7. Prior chemotherapy for recurrent or metastatic endometrial cancer is permitted.
8. Patients must have measurable disease as defined by the presence of bidimensionally measurable lesions with clearly defined margins on x-ray, scan (CT or MRI) or physical exam.
9. Adequate bone marrow reserve: granulocyte count > 1.5 x 109/L, hemoglobin > 9 g/dL (transfusion-independent) and platelets > 100,000 K/UL.
10. Adequate liver and renal function as defined as: total bilirubin value < 1.5 mg/dL; SGPT < 2x the upper limit of normal or < 5x the upper limit of normal when liver metastases are present; serum creatinine value of < 1.8 mg/dL. All qualifying laboratory parameters must be determined within one week of first treatment.
11. Patient compliance and geographic proximity that allows adequate follow-up.
12. Signed informed consent.

Exclusion Criteria:

1. Patients with serous or clear cell carcinomas of the endometrium.
2. Patients whose tumor is known to be PR negative.
3. Uncontrolled hypercalcemia.
4. Patients taking phenytoin, phenobarbital or carbamazepine.
5. Known predisposition to thromboembolic disorder, which in the investigator's judgment would put the patient at unacceptable risk for thromboembolic complications.
6. Patients who have received treatment for brain metastases may be enrolled provided they have remained stable for at least 6 months after surgery or radiation.
7. Women taking estrogen, progestin or antiprogestins. Patients taking these drugs must have discontinued their use at least 3 weeks prior to beginning treatment with Mifepristone.
8. History of other malignancy (except adequately treated non-melanomatous carcinoma of the skin or cervical carcinoma in situ) unless in complete remission and off all therapy for that disease for a minimum of 5 years.
9. Use of any chemotherapy or investigational agent within 3 weeks prior to taking study drug.
10. Concurrent serious infection.
11. Patients with serious intercurrent medical illness.
12. Serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator).
13. Patients whom absorption of drugs is likely to be impaired due to either concomitant medications or prior surgery.
14. Overt psychosis or mental disability or otherwise incompetent to give informed consent.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2001-09; Primary Completion 2007-10 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Overall Response | With each 4 week cycle, follow up 2 years
  Overall Response = Complete and Partial Responses

CONTACTS AND LOCATIONS:
Overall Officials: Lois M. Ramondetta, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org